CLINICAL TRIAL: NCT06288321
Title: Randomized Controlled Trial Comparing the Efficacy and Safety of Mydriatic Microdrops Over Standard Dose Mydriatics for Pupil Dilation in Retinopathy of Prematurity Examination
Brief Title: A Study Investigating Whether Low Dose Eyedrops for Pupil Dilation is as Effective and Safe as Standard Dose Eyedrops in Examination for Retinopathy of Prematurity.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lu Evelyn Ruoyun, Doctor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: UW22221
Record Dates: First submitted 2024-02-18; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of prematurity; Preterm; Retinopathy of prematurity screening; Microdrops; Mydrin P; Mydriatics
MeSH Terms: conditions — Retinopathy of Prematurity; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Mydrin-P Group (Placebo Comparator): Subjects allocated to the Standard Mydrin P group will receive standard Mydrin-P (0.5% tropicamide / 0.5% phenylephrine HCl) which is the standard eyedrops used for dilation of pupil before retinopathy of prematurity examination.
  Interventions: Drug: Standard Mydrin-P
- Microdrop group (Experimental): Those allocated to the microdrop group will receive microdrop Mydrin-P for pupil dilation before retinopathy of prematurity exam.
  Interventions: Drug: Microdrop Mydrin-P

INTERVENTIONS:
Drug: Microdrop Mydrin-P — Microdrop Mydrin-P consists of around one third of the standard Mydrin-P drop size. Drop volume measurement was performed using a precision weight scale (Sartorius) with accuracy up to 0.001g. The microdrop administration was conducted via attachment of a 16 gauge needle to a 1ml syringe.
  Arms: Microdrop group
Drug: Standard Mydrin-P — Standard Mydrin-P is the standard mydriatic used for retinopathy of prematurity exam as per our local usual practice.
  Arms: Standard Mydrin-P Group

SUMMARY:
A prospective, randomized controlled study was conducted from August, 2022 to March, 2023 in the neonatal intensive care unit in Queen Mary Hospital, Hong Kong. The aim of this study was to determine whether microdrops Mydrin-P demonstrates similar efficacy as standard Mydrin -P eyedrops applied to neonates undergoing retinopathy of prematurity (ROP) screening exams, also to ascertain the optimal time for eye examination after administration of mydriatics and assess whether the cardiovascular, respiratory and gastrointestinal adverse effects differ between microdrops and standard dose Mydrin-P.

Preterm infants were randomized to receive either the standard Mydrin-P eyedrops or the mydriatic microdrops which contained around one-third of the standard Mydrin-P dosage. The primary outcome measured whether a successful ROP examination was conducted. Secondary outcomes included pupil diameters at baselines, 30 minutes, 60 minutes, 120 minutes after eyedrops instillation and at the time of ROP exam as well as adverse effects followed by the mydriatics administration.

A total of 18 patients were enrolled in this study with total 46 episodes of ROP recorded. All episodes with microdrops instillation led to successful ROP exams. There was no statistically significant difference between standard eyedrops and microdrops in determining the success of ROP exam (p=0.233). Mean pupil diameter did not differ between the microdrops and standard eyedrops group. At the time of ROP exam, the mean pupil diameter was 5.47mm in the standard eyedrops group and 5.73mm in the microdrops group. The optimal time for ROP exam was 60 minutes to 120 minutes after first dose of mydriatic. Also there was no difference in the occurrence of systemic side effects when compared to standard Mydrin P drops.

Hence the study concluded that microdrops have similar efficacy and safety profile compared to standard Mydrin-P eyedrops.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with estimated gestational age (EGA) at birth ≤32 weeks
* Neonates with birth weight ≤1500g

Exclusion Criteria:

* Neonates with severe clinical condition with unstable vital signs
* Neonates with congenital anomalies, syndromic disease
* Neonates with ophthalmological conditions such as eye infections, congenital eye anomalies, trauma
* Neonates with conditions that are contraindicated to mydriatic use

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Successfulness of a ROP exam | From the start of pupil dilation to pupil examination which is around 2 to 3 hours
  Primary outcome of the study was whether the ROP screening was successfully performed or not without additional eyedrops defined by the ophthalmologist conducting the exam.

SECONDARY OUTCOMES:
Pupil diameters | From start of pupil dilation (baseline) to 120 minutes after pupil dilation, total time is 120 minutes.
  Pupil diameter (in millimetres, mm) was documented at baseline (before eyedrops are applied, T0), 30 minutes from first dose of eyedrop (T30), 60 minutes from first dose of eyedrop (T60), 120 minutes from first dose of eyedrop (T120) and at time of ROP exam (TROP). Two measurements were taken during each time, one by visual assessment, another one by pupillometer measurement.
Heart rate | From start of pupil dilation (baseline) to 120 minutes after pupil dilation, total time is 120 minutes.
  Heart rate at baseline (before eyedrops are applied, T0), 30 minutes from first dose of eyedrop (T30), 60 minutes from first dose of eyedrop (T60), 120 minutes from first dose of eyedrop (T120) and at time of ROP exam (TROP) were captured.
Blood pressure | From start of pupil dilation (baseline) to 120 minutes after pupil dilation, total time is 120 minutes.
  Blood pressure at baseline (before eyedrops are applied, T0), 30 minutes from first dose of eyedrop (T30), 60 minutes from first dose of eyedrop (T60), 120 minutes from first dose of eyedrop (T120) and at time of ROP exam (TROP) were captured.
Oxygen saturation | From start of pupil dilation (baseline) to 120 minutes after pupil dilation, total time is 120 minutes.
  Oxygen saturation at baseline (before eyedrops are applied, T0), 30 minutes from first dose of eyedrop (T30), 60 minutes from first dose of eyedrop (T60), 120 minutes from first dose of eyedrop (T120) and at time of ROP exam (TROP) were captured.
Oxygen requirement | From start of pupil dilation (baseline) to 120 minutes after pupil dilation, total time is 120 minutes.
  Oxygen requirement at baseline (before eyedrops are applied, T0), 30 minutes from first dose of eyedrop (T30), 60 minutes from first dose of eyedrop (T60), 120 minutes from first dose of eyedrop (T120) and at time of ROP exam (TROP) were captured.
Episodes of vomiting | From start of pupil dilation (baseline) to 24 hours after pupil dilation, total time is 24 hours.
  Episodes of vomiting were documented in the 24 hours after eyedrops administration and compared to the baseline which is the past 24 hours prior to the eyedrops exposure
Volume of gastric residuals | From start of pupil dilation (baseline) to 24 hours after pupil dilation, total time is 24 hours.
  Volume of gastric residuals were documented in the 24 hours after eyedrops administration and compared to the baseline which is the past 24 hours prior to the eyedrops exposure
Episodes of apnoea | From start of pupil dilation (baseline) to 24 hours after pupil dilation, total time is 24 hours.
  Episodes of apnoea were documented in the 24 hours after eyedrops administration and compared to the baseline which is the past 24 hours prior to the eyedrops exposure
Episodes of periorbital blanching | From start of pupil dilation (baseline) to 24 hours after pupil dilation, total time is 24 hours.
  Episodes of periorbital blanching were documented in the 24 hours after eyedrops administration and compared to the baseline which is the past 24 hours prior to the eyedrops exposure

CONTACTS AND LOCATIONS:
Overall Officials: Khair Jalal, Study Chair — Department of Paediatrics and Adolescent Medicine, Queen Mary Hospital
Locations (1):
- Department of Paediatrics and Adolescent Medicine, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT06288321/Prot_000.pdf